CLINICAL TRIAL: NCT05192694
Title: Evaluation of Fapi-pet in Prostate Cancer
Acronym: FAPIPETPCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Antti Rannikko, Assistant professor, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUS/2997/2021
Record Dates: First submitted 2021-12-07; First posted 2022-01-14 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: PET; PSMA; FAP; radical prostatectomy; novel antiandrogen; enzalutamide; apalutamide; FAPi; exosome
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Exploratory prospective cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FAPI PET (Other): Prospective single arm cohort
  Interventions: Procedure: Computed tomography

INTERVENTIONS:
Procedure: Computed tomography — Positron Emission Tomography
  Other Names: 68-Ga-FAPI-4 PET/CT

SUMMARY:
The investigators explore the biodistribution of FAPI-PET expression in primary high-risk prostate cancer in men undergoing RALP and eLND and in men with metastatic PCa about to start next generation antiandrogen.

DETAILED DESCRIPTION:
This is an exploratory cohort study comprised of men with clinically localized or locally advanced high-risk prostate cancer (GG 3-5, cT2-cT3, Nx, M0) managed by RALP and eLND and men with metastatic (mHSPC or mCRPC) prostate cancer scheduled to start NHT along clinical care pathway (e.g., apalutamide, enzalutamide) at HUS Helsinki University Hospital and Helsinki University, Finland.

Men identified along routine clinical care as candidates for the study will be asked to consent.

Once consented, patients will undergo PSMA-PET imaging instead of conventional imaging (CT and bone scan) and experimental FAPI-PET imaging. Furthermore, biomarker samples will be obtained before and after treatment (surgery or novel antiandrogen) and surgical specimen will be processed for routine pathological evaluation and multiplex IHC studies. Serum samples will be tested for PCa biomarkers (e.g., PSA, NSE, CgA) and cfDNA. Urine will be processed and extracellular vesicles (exosomes) isolated and markers of reactive stroma will be sought for.

Radical prostatectomy and novel hormonal treatment will be done according to current recommendations and guidelines in Finland.

Postoperatively, patients will be followed with PSA every six months. Biochemical recurrence will be set at PSA of 0.2 ug/l or higher.

ELIGIBILITY:
Inclusion Criteria:

Men scheduled for radical prostatectomy

* Age over 18 years
* GG 3-5, cT2-cT3, Nx, M0 prostate cancer
* no contraindication to PSMA - or FAPI-PET
* willing to undergo study related procedures (imaging and laboratory tests) Men scheduled for novel antiandrogen
* Age over 18 years
* GG2-5, cT2-4, N0-1, M1
* hormone sensitive or castration resistant prostate cancer

Exclusion Criteria:

* Not willing or capable to undergo study related procedures

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value on a lesion level | through study completion, an average of 1 year
  Positive predictive value of FAPI-PET on a lesion level using histopathology or confirmatory imaging as ground truth

SECONDARY OUTCOMES:
Positive predictive value on a patient level | through study completion, an average of 1 year
  Positive predictive value of FAPI-PET on a patient level using histopathology or confirmatory imaging as ground truth
To assess the biodistribution of FAPI PET signal in comparison to PSMA-PET signal | through study completion, an average of 1 year
  To explore and compare the biodistribution and signal level of FAPI-PET and PSMA-PET
To assess the biodistribution of FAPI and PSMA PET signal in comparison to histology | through study completion, an average of 1 year
  To explore the biodistribution and signal level of FAP-PET and PSMA-PET in correlation to reference histology (lesion volume and grade in radical prostatectomy specimen and lymphadenectomy specimen)
To assess the biodistribution of FAPI and PSMA PET signal in comparison to immunohistochemistry | through study completion, an average of 1 year
  To explore the biodistribution and signal level of FAPI-PET and PSMA-PET in correlation to tissue protein levels of:
  1. FAP and PSMA
  2. Markers of reactive stroma and CAFs
  3. Neuregulin-1
  4. Androgen receptor signalling pathway
To assess the biodistribution of FAPI and PSMA PET signal in comparison to biomarkers in "wet" samples | through study completion, an average of 1 year
  To correlate FAPI-PET and PSMA-PET biodistribution and signal level to:
  1. Postoperative serum biomarker levels (e.g., PSA, afos)
  2. cfDNA/RNA levels in peripheral blood
  3. Urinary exosome status for markers of reactive stroma
  4. Biochemical recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Antti S Rannikko, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol
Time Frame: during the study
Access Criteria: publically available at the study group web site once study starts.
URL: http://hucc.fi

REFERENCES:
- See also: study group website — http://www.hucc.fi